CLINICAL TRIAL: NCT01499069
Title: Urinary NGF, PGE2 and ATP: Potential Biomarkers for Diagnosis and Prediction of Treatment Efficacy in Overactive Bladder Patients
Brief Title: Urinary Nerve Growth Factor (NGF), Prostaglandin E2 (PGE2)and Adenosine Triphosphate (ATP): Potential Biomarkers in Overactive Bladder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Biomedical Research Institute (Unknown)
Responsible Party: Principal Investigator, KYU-SUNG LEE, Professor of Urology, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2009-09-036
Record Dates: First submitted 2011-05-24; First posted 2011-12-26 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine; Solifenacin Succinate; propiverine; trospium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antimuscarinic agents (Experimental)
  Interventions: Drug: Oxybutinin, Fesoterodine, Solifenacin, Propiverin, Trospium

INTERVENTIONS:
Drug: Oxybutinin, Fesoterodine, Solifenacin, Propiverin, Trospium — Dosage and frequency can be adjusted according to the patients' symptoms based on the instruction for administration .
  Duration; 3 or 6 months

SUMMARY:
Nerve growth factor (NGF), prostaglandin E2 (PGE2)and adenosine triphosphate (ATP) levels in urine were reported to increase in patients with overactive bladder (OAB). Also, administration of the anti-muscarinic agent was reported to decrease urinary NGF and ATP.

The investigators aimed to explore the value of the urinary NGF, PGE2 and ATP as biomarker for predicting the treatment responsiveness and symptom relapse in OAB patients. So, the patients can be categorized into responder or non- responder and relapse or non-relapse groups. Ultimately, they can receive individualized treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or over 18 years who had no history of antimuscarinic treatment or stopped antimuscarinics at least 3 months prior to the screening visit
* Verified by 3-day bladder diary as below

  * Urgency episode of 2 or over 2 times/24 hours (defined as a level of 3 to 5 in a 5 point urgency scale at baseline)
  * Urinary frequency of 8 or over 8 times/24 hours
* Symptom duration of 3 or over 3 months.
* Ability and willingness to correctly complete the micturition diary and questionnaire
* Capable of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

* Clinically significant stress incontinence as determined by the investigators and confirmed for female patients by a cough provocation test.
* Significant hepatic or renal disease, defined as having twice the upper limit of the reference ranges for serum concentrations of aspartate aminotransferase (AST [SGOT]), alanine aminotransferase (ALT [SGPT]), alkaline phosphatase or creatinine
* Any condition that is a contraindication for anticholinergic treatment, including uncontrolled narrow-angled glaucoma, urinary retention or gastric retention
* Symptomatic acute urinary tract infection (UTI) during the run-in period
* Recurrent UTIs defined as having been treated for symptomatic UTIs > 4 times in the last year
* Diagnosed or suspected interstitial cystitis
* Uninvestigated hematuria or hematuria secondary to malignant disease.
* Clinically significant bladder outlet obstruction defined by clinical symptoms and investigator's opinion according to local standard of care
* Patients with marked cystocele or other clinically significant pelvic prolapse.
* Treatment within the 14 days preceding randomization, or expected to initiate treatment during the study with:

  * Any anticholinergic drugs other than randomized trial drug
  * Any drug treatment for overactive bladder. Estrogen treatment started more than 2 months prior to inclusion is allowed.
* On an unstable dosage of any drug with anticholinergic side effects, or expected to start such treatment during the study
* Receipt of any electrostimulation or bladder training within the 14 days before randomization, or expected to start such treatment during the study
* An indwelling catheter or practicing intermittent self-catheterization
* Use of any investigational drug within 2 months preceding the start of the study
* Patients with chronic constipation or history of severe constipation
* Pregnant or nursing women
* Sexually active females of childbearing potential not using reliable contraception for at least 1 month prior to study start and not agreeing to use such methods during the entire study period and for at least 1 month thereafter. Reliable contraceptive methods are defined as intrauterine devices (IUDs), combination type contraceptive pills, hormonal implants, double barrier method, injectable contraceptives and surgical procedures (tubal ligation or vasectomy).
* Patients who have bladder cancer or prostate cancer
* Treatment with potent CYP3A4 inhibitors, such as cyclosporine, vinblastine, macrolide antibiotics (e.g. erythromycin, clarithromycin, azithromycin) or antifungal agents (e.g. ketoconazole, itraconazole, micronazole).
* Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2010-02; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
NGF/creatinine, PGE2/creatinine and ATP/creatinine level at pre-treatment and post-treatment of overactive bladder patients. | 3 months after antimuscarinics medication (if, the improvement of symptoms meet the criteria of treatment completion at 3 months of medicaion) and 3 months after medication completion

SECONDARY OUTCOMES:
NGF/creatinine, PGE2/creatinine and ATP/creatinine level at pre-treatment and post-treatment of overactive bladder patients. | 1 month after antimuscarinics medication and 1 months after medication completion
NGF/creatinine, PGE2/creatinine and ATP/creatinine level at pre-treatment and post-treatment of overactive bladder patients. | 4 and 6 months after antimuscarinics medication (if, the improvement of symptoms do not met the criteria of treatment completion at 3 months of medicaion)

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea